CLINICAL TRIAL: NCT01281410
Title: Effectiveness of an Inspiratory Muscle Training in Patients Receiving Allogenic Stem Cell Transplantation
Brief Title: Inspiratory Muscle Training in Patients Receiving Allogenic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elisabethinen Hospital (Other)
Responsible Party: Ursula Raschhofer,MSc, Elisabethinen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK 462
Record Dates: First submitted 2011-01-18; First posted 2011-01-24 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2010-11

CONDITIONS: Inspiratory Muscle Training; Stem Cell Transplantation; Respiratory Muscle Training
Keywords: respiratory muscles; hematopoetic stem cell transplantation; inspiratory muscle training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard physiotherapy (No Intervention): Standard Physiotherapy without Inspiratory Muscle Training
- Inspiratory muscle training (Experimental): Inspiratory muscle training with a device named Respifit in addition to the usual physiotherapy program
  Interventions: Procedure: Inspiratory Muscle Training; Other: inspiratory muscle training

INTERVENTIONS:
Procedure: Inspiratory Muscle Training — Inspiratory Muscle Training with Respifit (5 times per week)
  Arms: Inspiratory muscle training
Other: inspiratory muscle training — Inspiratory muscle training with a device named Respifit for patients receiving a hematopoetic stem cell transplantation (till 30 days after their transplantation)
  Arms: Inspiratory muscle training

SUMMARY:
The study is a monocentric, controlled randomized trial. Its an interventional method study. There is a control and an interventional group. The interventional group is receiving a specific inspiratory muscle training with "Respifit" (special device for inspiratory muscle training) during the first 30 days after allogenic stem cell transplantation.

The investigators want to show that the training group gets stronger inspiratory muscles. The investigators measure the change of PIMAX values and MVV values.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving allogenic stem cell transplantation
* Age 17 - 80 years old
* Informed consent

Exclusion Criteria:

* Actual pneumonia at the beginning of the trial
* Impaired vision
* Patient is not able to handle "Respifit"

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Change of PI max-value from baseline at 30 days after stem cell transplantation | baseline and 30 days after stem cell transplantation
  max strength of the inspiratory muscles
Change of MVV-value from baseline at 30 days after transplantation | baseline and 30 days after stem cell transplantation
  max voluntary volume for Inspiratory muscle endurance

SECONDARY OUTCOMES:
inpatient days | from baseline to maximal 60 days after stem cell transplantation
Incidence of pneumonia | from baseline to 30 days after stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Hanns Hauser, MD, Study Chair — Elisabethinen Hospital
Locations (1):
- Elisabethinen Hospital, Linz, Austria